CLINICAL TRIAL: NCT05072743
Title: Improvement in Sleep Symptomatology and Neurocognitive Function Using Photobiomodulation in Post-Concussion Patients With Sleep-Wake Disturbances
Brief Title: Improvement in Sleep Symptomatology and Neurocognitive Function Using Photobiomodulation in Post-Concussion Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Zitney (Other)
Collaborators: Meditech Rehabilitation Centre (Other)
Responsible Party: Sponsor-Investigator, Michael Zitney, Medical Director, Meditech Rehabilitation Centre
Organization: Meditech Rehabilitation Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFX2
Record Dates: First submitted 2021-09-17; First posted 2021-10-11 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Post-Concussion Syndrome; Sleep Disorder
Keywords: Post-Concussion Syndrome; Photobiomodulation; Sleep Disorder
MeSH Terms: conditions — Post-Concussion Syndrome; Sleep Wake Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-Concussion Patients with Non-Apneic Sleep Disorder (Experimental): Patients will be treated with PBMT using the BIOFLEX® DUO+ system that utilizes a Light Emitting Diode (LED) array pad followed by laser probes. Both delivery methods will be applied to the cervical spine and will entail the use of red light at 660 nm wavelength and near-infrared light at 830-840 nm wavelength. Treatment is provided twice per week for 6 weeks for a total of 12 treatments utilizing Health Canada approved device specific protocol guidelines for the treatment of the cervical spine soft tissue injuries.
  Interventions: Device: Photobiomodulation Therapy

INTERVENTIONS:
Device: Photobiomodulation Therapy — PBMT will be applied to the cervical spine using the BIOFLEX® DUO+ system that utilizes a Light Emitting Diode (LED) array pad followed by laser probes. Both delivery methods will be applied to the cervical spine and will entail the use of red light at 660 nm wavelength and near-infrared light at 830-840 nm wavelength. Treatment is provided twice per week for 6 weeks for a total of 12 treatments utilizing Health Canada approved device specific protocol guidelines for the treatment of the cervical spine soft tissue injuries.
  Other Names: Low Level Laser Therapy

SUMMARY:
The emphasis on this study is to review the use of PBMT as a potential treatment modality to improve both sleep symptoms and consequent neuropsychological functions affected by sleep disturbances in a cohort of post-mTBI patients with sleep issues not secondary to sleep apnea.

DETAILED DESCRIPTION:
Concussion or mild traumatic brain injury (mTBI) is an acute neurophysiological event related to blunt impact applied to the head and/or neck due to sudden acceleration, deceleration or rotational forces. It can happen due to motor vehicle accidents, sport or recreational injury, falls, workplace injury or assault. mTBI can be differentiated from moderate and severe traumatic brain injuries by having negative imaging or laboratory results and a Glasgow Coma Scale (GCS) score of 13-15. Current treatment modalities for the various symptoms associated with mTBI are mostly supportive: pain medication, antidepressants, psychotherapy, physiotherapy, vision therapy and referral to sleep clinics.

mTBI symptoms are usually divided into four groups: cognitive symptoms, physical symptoms, emotional symptoms and sleep symptoms. Although most of these symptoms resolve or improve with or without treatment within 3 months following injury there is a significant population of post-mTBI patients who continue to suffer from symptoms 3 months to years after their injury. Previously called Post-Concussive Syndrome (PCS) most groups now classify PCS as a neurological disorder with persistent post-concussive symptoms. Insufficient and disturbed sleep are reported by half of all patients and are among the most common complaints following mTBI, and can develop during the early to chronic post-mTBI phases. Various sleep abnormalities, including post-TBI insomnia, hypersomnia, and sleep apnea are frequently observed. Most cases of sleep symptoms associated with mTBI that are diagnosed during sleep studies tend to be apnea related, although the cause of this is still unknown. Sleep apnea can be obstructive or central sleep apnea, but both types tend to respond well to Continuous Positive Airway Pressure. For other types of non-apneic sleep related symptoms post mTBI though, treatment can vary from Cognitive Behavioural Therapy (CBT) to various sleep medications. However, it is noted that despite an improvement in objective sleep symptoms with conventional approaches to patients with mTBI, there continues to be a lack of improvement in terms of subjective sleepiness or neuropsychological functions.

Photobiomodulation therapy (PBMT) is an innovative modality for the stimulation of neural activity in order to improve brain function and is currently under investigation as a treatment for several diverse neurological disorders, including concussions. Noted among the effects of PBMT among post-mTBI patients in our clinic is a subjective improvement in sleep, sometimes described by patients as "the best sleep they've ever had." Our emphasis on this study is to review the use of PBMT as a potential treatment modality to improve both sleep symptoms and consequent neuropsychological functions affected by their sleep disturbances in a cohort of post-mTBI patients with sleep issues not secondary to sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-70 years clinically diagnosed with a mTBI diagnosed between 3 to 24 months from presentation complaining of sleep disturbance.
* Underwent an overnight sleep study PSG within the previous year and diagnosed with a primary sleep disorder and in which there has been symptom development suggesting another co-morbid sleep disorder, or an established diagnosis of a sleep disorder other than a sleep related breathing disorder who have significant symptom progression or non-response to therapy.
* Documentation of a history of a qualifying mTBI within 3 to 24 months of traumatic incident and/or diagnosis with persistent symptomatology after 3 months. For reference, International Classification of Diseases, Tenth Revision (ICD-10) clinical criteria for Post Concussive Syndrome (PCS) require a history of TBI and the presence of three or more of the following eight symptoms: 1) headache, 2) dizziness, 3) fatigue, 4) irritability, 5) insomnia, 6) concentration or 7) memory difficulty, and 8) intolerance of stress, emotion, or alcohol4.

Exclusion Criteria:

* Any positive cranial findings on imaging studies
* A current diagnosis of neuropsychiatric co-morbidity including severe anxiety (or score of ≥15 on the GAD-7), severe depression (or score of ≥20 on the PHQ-9), schizophrenia or bipolar disorder.
* A family history of neuropsychiatric conditions
* Any additional diagnoses compounding the diagnosis of a mTBI.
* Currently undergoing CBT.
* Currently taking any medication for the purpose of improving sleep including medical and recreational cannabis, barbiturates, benzodiazepines, antidepressants, antihistamines, melatonin or other natural supplements.
* Currently undergoing any alternative or complementary medical procedure, i.e. acupuncture, hypnosis, homeopathy, etc.
* Pregnancy
* Malignant growth in the neck and cranium
* Taking any photosensitizing medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Statistically significant changes in the Epsworth Sleepiness Scale (ESS) scores from baseline and at 4 weeks | Baseline, 4 weeks
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Statistically significant changes in the Epsworth Sleepiness Scale (ESS) scores from baseline and at 8 weeks | Baseline, 8 weeks
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Statistically significant changes in the Epsworth Sleepiness Scale (ESS) scores from baseline and at 12 weeks | Baseline, 12 weeks
  The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Statistically significant changes in the Insomnia Severity Index (ISI) scores from baseline and at 4 weeks | Baseline, 4 weeks
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Statistically significant changes in the Insomnia Severity Index (ISI) scores from baseline and at 8 weeks | Baseline, 8 weeks
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Statistically significant changes in the Insomnia Severity Index (ISI) scores from baseline and at 12 weeks | Baseline, 12 weeks
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Statistically significant changes in the total duration (in total minutes) of Stage 3 Non Rapid Eye Movement (NREM) or N3 sleep during Type 1 overnight Polysomnography (OSG) from Baseline and at 8 weeks. | Baseline, 8 weeks
  Overnight measurement of sleep stage duration in minutes utilizing 3 studies: electroencephalography (EEG), electrooculography (EOG), and surface electromyography (EMG). Other parameters that may also be monitored to measure sleep stage duration include the following: Electrocardiography, Pulse oximetry, Respiratory effort (thoracic and abdominal), End tidal or transcutaneous Carbon Dioxide (CO2), Sound recordings to measure snoring, Surface EMG monitoring of limb muscles (to detect limb movements, periodic or other). These studies are consolidated by a sleep physician to determine and identify each sleep stage in minutes. Only data regarding the duration in minutes as identified by the sleep physician will be collected.
Statistically significant changes in the total duration (in total minutes) of Stage 4 Rapid Eye Movement (REM) sleep during Type 1 overnight Polysomnography (OSG) from Baseline and at 8 weeks | Baseline, 8 weeks
  Overnight measurement of sleep stage duration in minutes utilizing 3 studies: electroencephalography (EEG), electrooculography (EOG), and surface electromyography (EMG). Other parameters that may also be monitored to measure sleep stage duration include the following: Electrocardiography, Pulse oximetry, Respiratory effort (thoracic and abdominal), End tidal or transcutaneous Carbon Dioxide (CO2), Sound recordings to measure snoring, Surface EMG monitoring of limb muscles (to detect limb movements, periodic or other). These studies are consolidated by a sleep physician to determine and identify each sleep stage in minutes. Only data regarding the duration in minutes as identified by the sleep physician will be collected.

SECONDARY OUTCOMES:
Statistically significant changes in the Functional Outcomes of Sleep Questionnaire (short version) (FOSQ-10) scores from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  The short 10-item version of the original 30 item FOSQ using selected items from each subscale and providing the same definition of sleepy and tired. Items for the FOSQ-10 are distributed among the same subscales as follows: 1) activity level (3 items), 2) vigilance (3 items), 3) intimacy and sexual relationships (1 item), 4) general productivity (2 items), and 5) social outcomes (1 item).
Statistically significant changes in the Motivation and Energy Inventory Short Form (MEI-SF) scores from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  The MEI-SF is AN 18-item scale created to assess fatigue and lassitude. The scale was initially developed for the purpose of evaluating interventions to improve motivation and energy in patients with depression, though with further evaluation, its clinical applications could be extended to other patient groups. The MEI assesses three factors: mental or cognitive energy, social motivation, and physical energy.
Statistically significant changes in the Rivermead Post-Concussion Symptoms Questionnaire (RPQ) scores from baseline | Baseline, 4 weeks, 8 weeks, 12 weeks
  RPQ is a self-report scale to measure the severity of post-concussive symptoms following a Traumatic Brain Injury (TBI). It is a 16-item self-report questionnaire that assesses the severity of 16 different PCS symptoms that typically follow TBI. Patients are asked to rate their symptoms before and after their injury and also to rate the severity of their symptoms in the last 24 h. Items follow a 5-point ordinal rating system where 0 = never experienced at all, 1 = no more of a problem, 2 = a mild problem, 3 = a moderate problem, and 4 = a severe problem. Thus total scores using the sum of all items can theoretically range from 0 to 64.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Lowe, MD, Principal Investigator — Meditech International; Michael Zitney, MD, Principal Investigator — MediTech International Inc.
Locations (1):
- Meditech Rehabilitation Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tator CH. Concussions and their consequences: current diagnosis, management and prevention. CMAJ. 2013 Aug 6;185(11):975-9. doi: 10.1503/cmaj.120039. Epub 2013 Jul 22. No abstract available. PMID 23877672
- [Background] Zemek R, Barrowman N, Freedman SB, Gravel J, Gagnon I, McGahern C, Aglipay M, Sangha G, Boutis K, Beer D, Craig W, Burns E, Farion KJ, Mikrogianakis A, Barlow K, Dubrovsky AS, Meeuwisse W, Gioia G, Meehan WP 3rd, Beauchamp MH, Kamil Y, Grool AM, Hoshizaki B, Anderson P, Brooks BL, Yeates KO, Vassilyadi M, Klassen T, Keightley M, Richer L, DeMatteo C, Osmond MH; Pediatric Emergency Research Canada (PERC) Concussion Team. Clinical Risk Score for Persistent Postconcussion Symptoms Among Children With Acute Concussion in the ED. JAMA. 2016 Mar 8;315(10):1014-25. doi: 10.1001/jama.2016.1203. PMID 26954410
- [Background] Ruff RM. Mild traumatic brain injury and neural recovery: rethinking the debate. NeuroRehabilitation. 2011;28(3):167-80. doi: 10.3233/NRE-2011-0646. PMID 21558623
- [Background] Mathias JL, Alvaro PK. Prevalence of sleep disturbances, disorders, and problems following traumatic brain injury: a meta-analysis. Sleep Med. 2012 Aug;13(7):898-905. doi: 10.1016/j.sleep.2012.04.006. Epub 2012 Jun 15. PMID 22705246
- [Background] Schreiber S, Barkai G, Gur-Hartman T, Peles E, Tov N, Dolberg OT, Pick CG. Long-lasting sleep patterns of adult patients with minor traumatic brain injury (mTBI) and non-mTBI subjects. Sleep Med. 2008 Jul;9(5):481-7. doi: 10.1016/j.sleep.2007.04.014. Epub 2007 Jul 16. PMID 17638592
- [Background] Castriotta RJ, Atanasov S, Wilde MC, Masel BE, Lai JM, Kuna ST. Treatment of sleep disorders after traumatic brain injury. J Clin Sleep Med. 2009 Apr 15;5(2):137-44. PMID 19968047
- [Background] Salehpour F, Mahmoudi J, Kamari F, Sadigh-Eteghad S, Rasta SH, Hamblin MR. Brain Photobiomodulation Therapy: a Narrative Review. Mol Neurobiol. 2018 Aug;55(8):6601-6636. doi: 10.1007/s12035-017-0852-4. Epub 2018 Jan 11. PMID 29327206
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chasens ER, Ratcliffe SJ, Weaver TE. Development of the FOSQ-10: a short version of the Functional Outcomes of Sleep Questionnaire. Sleep. 2009 Jul;32(7):915-9. doi: 10.1093/sleep/32.7.915. PMID 19639754
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320